CLINICAL TRIAL: NCT00938860
Title: A Multi-center, Randomized, Open Label, Controlled Study to Compare the Sustained Virological Response During Treatment With Neoral or Tacrolimus in Maintenance Liver Transplant Recipients Treated With Pegylated Interferon and Ribavirin for Recurrent Hepatitis C
Brief Title: Sustained Virological Response (SVR) to Antiviral Treatment of Liver Transplant Recipients With Recurrent Hepatitis C
Acronym: SUSTAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLO400A2430; 2009-010806-12
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis C; Liver Transplantation
Keywords: Hepatitis C; liver transplantation; anti-viral therapy
MeSH Terms: conditions — Hepatitis C | interventions — Cyclosporine; Tacrolimus

ARMS (2):
- Neoral (Experimental): Neoral capsules bid, Doses were to be adjusted as necessary to achieve and maintain recommended C0 (monitoring of trough levels) or C2 concentration 2 hours post dosing) target ranges
  Interventions: Drug: cyclosporin (Neoral)
- tacrolimus (Active Comparator): Tacrolimus capsules bid, doses were adjusted as necessary to achieve and maintain recommended C0 target ranges.
  Interventions: Drug: tacrolimus (Prograf)

INTERVENTIONS:
Drug: cyclosporin (Neoral) — Neoral capsules bid, Doses were to be adjusted as necessary to achieve and maintain recommended C0 (monitoring of trough levels) or C2 concentration 2 hours post dosing) target ranges
  Arms: Neoral
Drug: tacrolimus (Prograf) — Tacrolimus capsules bid, doses were adjusted as necessary to achieve and maintain recommended C0 target ranges.
  Arms: tacrolimus

SUMMARY:
This study will assess the rates of Sustained Virological Response following anti-viral therapy with Peg-Interferon plus Ribavirin in patients that have been liver transplanted with recurrent Hepatitis C and treated with Neoral or tacrolimus.

ELIGIBILITY:
Inclusion criteria:

* Liver transplantation performed at least 6 months and up to 5 years prior randomization and due to HCV cirrhosis, with or without pre-transplant hepatocellular carcinoma (HCC) within Milan or UCSF criteria
* Immunosuppresive regimen based on tacrolimus b.i.d.- (twice or once daily) for at least 6 months prior randomization
* Diagnosis of HCV genotypes 1 or 4 infection prior to transplantationconfirmed at screening
* Indication of treatment with Peg-IFN and ribavirin due to histological evidence of chronic HCV infection defined as a fibrosis stage equal or greater than 1 using the Ishak-Knodell scoring system (IK ≥1) in a liver biopsy performed at screening or up to 4 months prior to randomization.

Exclusion criteria:

* Serum creatinine >150 μmol/L (1.6 7 mg/dL) or eGFR < 50 ml/min (4-variable Modification of Diet in Renal Disease [MDRD Cockcroft-Gault formula])
* Multi-organ transplant recipients
* Recent episode of steroid-treated acute rejection (AR) within 3 months prior to randomization, or >1 episode of steroid-treated AR in the last 6 months, or any number of steroid-resistant AR episodes in the last 6 months including evidence of chronic rejection or ductopenia
* Evidence of conditions that could cause graft dysfunction other than HCV infection
* Patients with signs of decompensated liver disease, defined as presence of ascites, variceal bleeding, encephalopathy or deteriorated hepatic synthetic function (albumin <3.5g/dL or, total direct bilirubin >1.5mg/dL or, INR >1.5)
* Co-infection with HIV or Hepatitis B (defined as HBsAg-positive) at screening
* Use of mTOR inhibitors (everolimus or sirolimus) in the 6 months prior to screening
* Antiviral treatment for HCV administered at any time after liver transplantation
* Patients on daily doses of corticosteroids higher than 5 mg/day
* Patients with fibrosing cholestatic hepatitis
* Patients with current diagnosis of malignancies, including lymphoproliferative disorders
* Patients with platelet count <70,000/mm3 or neutrophiles <1,500/mm3
* History of HCC outside Milan criteria based on radiology or UCSF criteria based on analysis of the explant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- United States (8):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Madison, Wisconsin
- Novartis Investigative Site, Brussels, Belgium
- Brazil (2):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Colombia (2):
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Bogotá
- France (6):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, München
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Udine, UD
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (4):
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
- Novartis Investigative Site, Zurich, Switzerland, Switzerland
- Novartis Investigative Site, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an 80 week multicenter randomized, open label, controlled study in adult HCVpositive maintenance liver transplant recipients. Patients were randomized at a 1.3:1 ratio to CsA and tacrolimus. Patients randomized to tacrolimus were maintained on treatment with tacrolimus, patients randomized to CsA were converted from tacrolimus to CsA
Groups:
- Neoral: Neoral® (cyclosporine for microemulsion), available as 10 mg, 25 mg, 50 mg and 100 mg soft gelatin capsules taken on a twice daily (b.i.d) schedule at 12-hour intervals, Doses were to be adjusted as necessary to achieve and maintain recommended C0 (monitoring of trough levels) or C2 concentration 2 hours post dosing) target ranges
- Tacrolimus: Prograf® (tacrolimus) provided as 0.5 mg, 1 mg and 5 mg capsules taken on a twice daily (b.i.d) schedule at 12-hour intervals. Doses were adjusted as necessary to achieve and maintain recommended C0 target ranges
Period: Overall Study
Arm/Group | Neoral | Tacrolimus
Started | 50 (Intent-to-Treat (ITT) population. ITT population consisted of all randomized patients) | 42
Efficacy Population | 40 | 41
Completed | 25 | 25
Not Completed | 25 | 17
Not completed — Adverse Event | 2 | 1
Not completed — Abnormal laboratory values | 2 | 2
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Lost to Follow-up | 4 | 4
Not completed — Administration problems | 2 | 0
Not completed — Death | 1 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population:
  The ITT population consisted of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Neoral | Tacrolimus | Total
Number analyzed (Participants) | 50 | 42 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (6.30) | 55.0 (6.84) | 54.6 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 41 | 34 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Sustained Virological Response (SVR) Following Treatment of Hepatitis C Virus (HCV) Infection With Peg-IFN and Ribavirin in Liver Transplanted Recipients on Maintenance Therapy With Neoral or Tacrolimus
Description: The achievement of SVR, defined as HCV RNA below limit of detection at the end of AV treatment, 24 weeks after end of AV treatment (W24 post). A dichotomous variable (SVR achieved: Yes/No) was computed. A patient was classified as non-responder (SVR not achieved) if HCV RNA was detectable at the completion of antiviral treatment, at W24post, or at any time between W24 and completion of antiviral treatment. The HCV RNA detection limit was <15 IU/ml (<1.18 log IU/ml)
Time Frame: Week 24
Population: The efficacy population was defined as a subset of the ITT population with sufficient compliance to the protocol procedures to allow meaningful conclusions. Patients were excluded from the Efficacy population in case of: Error in treatment assignment, if the randomized study medication was not initiated, antiviral therapy was not initiated
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 20 | 23
Participants | 12 | 10

2. Secondary Outcome: Number of Events of the Composite Endpoint of Biopsy Proven Acute Rejections (BPAR), Death or Graft Loss and of the Individual Components
Description: Efficacy failure (biopsy proven acute rejection (BPAR), graft loss, or death
Time Frame: Week 80
Population: Intent-to-Treat (ITT) population: The ITT population consisted of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Number; unit: Number of events
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 50 | 42
Number of events
  BPAR, graft loss, or death | 2 | 1
  BPAR | 1 | 0
  Graft loss or death | 1 | 1
  Death | 1 | 1

3. Secondary Outcome: Number of Participants With Fibrosis Progression (Increase in Ishak-Knodell (IK) Score by at Least One Point From the Baseline)
Description: Ishak-Knodell Score: 0=No fibrosis; 01=Fibrous expansion of some portal areas, with or without short fibrous septa; 02=Fibrous expansion of most portal areas, with or without short fibrous septa; 03=Fibrous expansion of most portal areas, with occasional portal to portal (P-P) bridging; 04=Fibrous expansion of portal areas, with marked bridging (portal to portal (P-P) as well as portal to central (P-C)); 05=Marked bridging (P-P and/or P-C) with occasional nodules (incomplete cirrhosis); 06=Cirrhosis, probable or definite, Participants showing an increase of Ishak Knodell fibrosis score by at least one level (increase of ≥1)
Time Frame: Week 80
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 13 | 17
Participants | 3 | 5

4. Secondary Outcome: Number of Participants of Rapid Viral Response (RVR)
Description: RVR defined as non-detectable HCV RNA 4 weeks after initiation of antiviral treatment. The HCV RNA detection limit was <15 IU/ml (<1.18 log IU/ml)
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 36 | 38
Participants | 4 | 5

5. Secondary Outcome: Number of Participants of Early Viral Response (EVR)
Description: EVR defined as non-detectable HCV RNA or a ≥2 logs reduction of HCV RNA at 12 weeks after initiation of antiviral treatment. The HCV RNA detection limit was <15 IU/ml (<1.18 log IU/ml)
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 31 | 36
Participants | 28 | 30

6. Secondary Outcome: Number of Participants for the End of Treatment Response (ETR)
Description: ETR defined as non-detectable HCV RNA at the completion of AV treatment. The HCV RNA detection limit was <15 IU/ml (<1.18 log IU/ml)
Time Frame: Week 80
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 35 | 39
Participants | 24 | 27

7. Secondary Outcome: Number of Participants of True Non-responder Rate
Description: Defined as failure to achieve at least a 2 log reduction of Hepatitis C virus (HCV) RNA. The HCV RNA detection limit was <15 IU/ml (<1.18 log IU/ml)
Time Frame: Week 80
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 40 | 41
Participants | 7 | 5

8. Secondary Outcome: Number of Participants for Relapse Rate
Description: Defined as reappearance of detectable Hepatitis C Virus (HCV) RNA at 24 weeks after completion of antiviral treatment when HCV RNA was undetectable at the end of treatment. The HCV RNA detection limit was <15 IU/ml (<1.18 log IU/ml)
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 23 | 21
Participants | 5 | 7

9. Secondary Outcome: Number of Participants With Dose Reduction or Discontinuation of Antiviral (AV) Therapy Due to Poor Tolerability at Any Time During the Study for Any Reason
Description: Defined as number of patients with dose reduction or discontinuation of AV therapy due to poor tolerability
Time Frame: Week 80
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Neoral | Tacrolimus
Number analyzed (Participants) | 40 | 41
Participants
  Neoral Antiviral treatment: Ribavirin | 25 | 0
  Neoral Antiviral treatment: Peg-IFN | 10 | 0
  Tacrolimus Antiviral treatment: Ribavirin | 0 | 23
  Tacrolimus Antiviral treatment: Peg-IFN | 0 | 11

ADVERSE EVENTS:
Arm/Group | Tacrolimus | Neoral
Serious Adverse Events (participants affected / at risk) | 17/42 | 18/50
Other Adverse Events (participants affected / at risk) | 41/42 | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=42) | Neoral (N=50)
Anaemia (Blood and lymphatic system disorders) | 5 | 6
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Exophthalmos (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver transplant rejection (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyoderma (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Urosepsis (Infections and infestations) | 0 | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=42) | Neoral (N=50)
Anaemia (Blood and lymphatic system disorders) | 28 | 27
Leukopenia (Blood and lymphatic system disorders) | 9 | 10
Neutropenia (Blood and lymphatic system disorders) | 14 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 11 | 9
Nausea (Gastrointestinal disorders) | 11 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 3
Asthenia (General disorders) | 10 | 7
Chills (General disorders) | 3 | 2
Fatigue (General disorders) | 13 | 12
Influenza like illness (General disorders) | 7 | 3
Irritability (General disorders) | 6 | 0
Oedema peripheral (General disorders) | 2 | 5
Pain (General disorders) | 0 | 3
Pyrexia (General disorders) | 5 | 8
Urinary tract infection (Infections and infestations) | 3 | 2
Haemoglobin decreased (Investigations) | 4 | 0
Neutrophil count decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 8 | 4
Headache (Nervous system disorders) | 7 | 8
Anxiety (Psychiatric disorders) | 2 | 3
Depression (Psychiatric disorders) | 4 | 7
Insomnia (Psychiatric disorders) | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety